CLINICAL TRIAL: NCT06103929
Title: Evaluation of Eating Difficulties Assessment Measures in Clinical Practice and in Epidemiological Surveys
Brief Title: Adult Eating Disorder Assessment Study
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: Leicestershire Partnership NHS Trust (Other); City, University of London (Other); National Centre for Social Research, London, UK (Unknown); University of London (Other)
Responsible Party: Principal Investigator, Sam Tromans, Associate Professor, University of Leicester
Other Study IDs: 0897
Record Dates: First submitted 2023-07-25; First posted 2023-10-27 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Eating Disorders
Keywords: Eating disorders; Adult psychiatry; Epidemiology; Calibration; Public health; Anorexia nervosa; Bulimia nervosa; Binge eating disorder
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults referred to eating disorder services: A cohort of adults referred to a specialist adult eating disorders service will be recruited. A stratified sample of patients will be approached about participating in the study, providing the study inclusion criteria are met, and their responsible clinician does not express concerns about their participation. All study participants will be assessed with the SCAN semi-structured interview (including version 2 of the SCAN, SCANv3s0, SCANv3s1, and SCANv3s9) and will also complete two self-completion measures, the EDE-QS and the SCOFF, randomly ordered. The SCAN items will be asked about in the context of the past 4 weeks and the directly preceding 11 months (i.e., the past year), unless otherwise stated. Additionally, a subset of study participants (n = 25) will be reassessed with the SCANv3s0, SCANv3s1, SCANv3s9, EDE-QS, and SCOFF, for test-retest reliability.

SUMMARY:
The hypothesis of the study is that low-cost self-completion questionnaires relating to eating disorder symptoms will predict the subsequent results of a detailed, semi-structured interview assessment of eating disorder symptoms that has been calibrated according to expert clinical diagnostic case thresholds. Eating disorders are recognised as a research priority among healthcare professionals, adults with lived experience, and their carers alike. There is a need for measurement methods that can reliably and systematically identify symptoms of common forms of eating disorder, including those fulfilling agreed diagnostic criteria for anorexia nervosa, bulimia nervosa, and binge-eating disorder. Effective diagnostic interview tools can facilitate early detection of eating disorders. To develop rules for determining whether diagnostic criteria for eating disorders are met, a study involving adults referred to specialist eating disorder services is required. In this study, assessments by eating disorder clinicians will be compared with researcher assessments using a semi-structured interview assessment, the Schedules for Clinical Assessment in Neuropsychiatry version 3 section 9 (SCANv3s9). The study population will consist of 100 adult patients referred to specialist eating disorder services, including patients whose referrals are accepted by these services, as well as those who are not. Clinical assessments and structured interview assessment findings will also be compared with those from widely used screening tools for eating disorders, the Eating Disorder Examination Questionnaire short-form and the SCOFF (Sick, Control, One, Fat, Food) questionnaire. The aim of this study is to evaluate the accuracy of the Eating Disorder Examination Questionnaire Short-Form (EDE-QS) and the SCOFF (Sick, Control, One, Fat, Food) questionnaire in adults referred to specialist eating disorder services, in a comparison with the Schedules for Clinical Assessment in Neuropsychiatry subsection on eating disorders and specialist NHS clinician assessments of the probability of eating disorder. This will help develop appropriate and accurate benchmarks for estimating the prevalence of eating disorder symptoms and clinical diagnoses, in adults referred to specialist eating disorder services, as well as the wider population (through combining the findings from this study with those of the community 2023 Adult Psychiatric Morbidity Survey).

DETAILED DESCRIPTION:
Study Analysis Plan

Work Package 1 (WP1) relates to assessment of the entire study clinical population (n = 100). For WP1, the threshold for diagnosis of common forms of eating disorders (anorexia nervosa, bulimia nervosa, binge-eating disorder, and any eating disorder) by clinicians will be used as the reference (criterion) standard, and 95% confidence intervals will be performed for all estimates. Receiver-operating characteristic (ROC) curves and areas under the curve (AUC) will be calculated for all measurement tools (SCANv3s9, EDE-QS, and SCOFF), with reference to the criterion standard, as well as sensitivity, specificity, positive predictive value, and negative predictive values for a range of cut-off scores for these tools. Additionally, correlation coefficients will be calculated with respect to SCANv3s9, EDE-QS, and SCOFF findings, relative to those of the reference standard.

To calibrate the SCANv3s9 interview, symptom findings from the researcher-assessed SCANv3s9 will be compared with NHS clinician's diagnostic thresholds. However, the research team may modify the SCANv3s9 diagnostic algorithms in the event that they diverge substantially from clinician judgment, an approach that has previously been employed when calibrating the Autism Diagnostic Observation Schedule (ADOS) against clinical opinion. Work Package 2 (WP2) relates to retesting of a subsample of the WP1 population (n = 25). For WP2, test-retest reliability will be assessed using Cohen's kappa coefficient (κ), as well as simple percentage agreement calculations.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 16 years or older (on the date of referral to specialist eating disorder services)
* Individuals referred to specialist adult eating disorder services during the study period

Exclusion Criteria:

* Patients under 16 years old and having not been referred to specialist eating disorder services.
* Patients with a clinical diagnosis of intellectual disability will be excluded on the basis that the SCAN is not intended for use in this patient group.
* Patients lacking capacity to consent to take part.
* Participants who lose capacity during their participation will be withdrawn from the study (with data collected up until the point of withdrawal being retained).
* Participants who are unable to understand written and verbal English.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Adults resident in the UK who have been referred to NHS Leicestershire Partnership Trust. The study aims to collect data on accepted referrals, which will represent the clinical population, and referrals not accepted into treatment which will represent people more likely to describe eating difficulties in community surveys.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The threshold on the questionnaires and SCAN examination output algorithm scores calibrated against the clinician diagnostic thresholds for eating disorder, taking account of the level of agreement between the questionnaires and SCAN | The WP1 SCAN interview battery (60-84 minutes)
  The SCAN assesses most forms of mental and neurodevelopmental disorders. SCANv3s9 is designed to measure eating disorder symptoms and the output numerical scores will be calibrated against clinician diagnostic thresholds for eating disorder (the criterion standard).
  The study will also ask about history of mental and physical health conditions

SECONDARY OUTCOMES:
The threshold on the EDE-QS examination output algorithm scores calibrated against the clinician diagnostic thresholds for eating disorder, taking account of the level of agreement between the EDE-QS and SCAN | The EDE-QS will take about 2.7 minutes to be completed
  The Eating Disorder Examination Short (EDE-QS) is a 12-item self-report questionnaire on eating disorder symptoms, and providing an overall numerical score. It showed high internal consistency, with reduced administration time.
The threshold on the SCOFF examination output algorithm scores calibrated against the clinician diagnostic thresholds for eating disorder, taking account of the level of agreement between the SCOFF and SCAN | The SCOFF (1.3 minutes) and basic demographic details form (3.7 minutes), completed by each participant
  The SCOFF questionnaire was used in the APMS survey in 2007, to screen for eating disorders. It is a 5-item measure, designed to detect eating disorders within a primary care setting.
  Please note that the respective measures of eating problems (SCAN, EDE-QS, and SCOFF) will be compared against the criterion standard (clinical diagnostic thresholds), but will not be aggregated to arrive at a singular reported value.
A retest comparison of findings from the SCAN among a subgroup of participants subject to repeated assessment | The reduced time of assessment due to repeat SCAN testing with SCANv3s0 and SCANv3s9, will take 20-28 minutes.
  A total of 25 participants will take part in WP2, all of whom will have previously participated in WP1. Most WP2 assessment will take place within 2-3 weeks of WP1 assessment. Although the WP2 research team assessments will also take place either in a clinical setting or the participant's home, as described in WP1, the participant in WP2 will be assessed by a different research team member than they were for WP1.
A retest comparison of findings from the EDE-QS among a subgroup of participants subject to repeated assessment | The EDE-QS will take about 2.7 minutes to be completed
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire, comprising fixed worded questions on eating disorder symptoms, and providing an overall score. A shortened version, the 12-item Eating Disorder Examination Short (EDE-QS) will be used
A retest comparison of findings from the SCOFF among a subgroup of participants subject to repeated assessment | The SCOFF (1.3 minutes) and basic demographic details form (3.7 minutes), completed by each participant
  The SCOFF questionnaire is a 5-item measure, designed to detect eating disorders within a primary care setting, with good validity when compared (for accuracy) with clinical diagnosis (DSM-IV).
  Please note that the respective measures of eating problems (SCAN, EDE-QS, and SCOFF) will be compared against the criterion standard (clinical diagnostic thresholds), but will not be aggregated to arrive at a singular reported value.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel J. Tromans, Principal Investigator — University of Leicester
Locations (1):
- Leicestershire Partnership NHS Trust, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the study, the data that support the findings of this study will be available to other researchers in deidentified form from the NHS Data Access Request Service or from another official data depository as yet to be determined.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: This will be made available starting January 2026
URL: https://le.ac.uk/people/sam-tromans

REFERENCES:
- [Background] Lord C, Risi S, Lambrecht L, Cook EH Jr, Leventhal BL, DiLavore PC, Pickles A, Rutter M. The autism diagnostic observation schedule-generic: a standard measure of social and communication deficits associated with the spectrum of autism. J Autism Dev Disord. 2000 Jun;30(3):205-23. PMID 11055457
- [Background] Brugha TS, McManus S, Smith J, Scott FJ, Meltzer H, Purdon S, Berney T, Tantam D, Robinson J, Radley J, Bankart J. Validating two survey methods for identifying cases of autism spectrum disorder among adults in the community. Psychol Med. 2012 Mar;42(3):647-56. doi: 10.1017/S0033291711001292. Epub 2011 Jul 29. PMID 21798110
- [Background] Fairburn CG, Cooper Z, O'Connor M. The eating disorder examination. 1993;6:1-8.
- [Background] McManus S, Bebbington PE, Jenkins R, Morgan Z, Brown L, Collinson D, Brugha T. Data Resource Profile: Adult Psychiatric Morbidity Survey (APMS). Int J Epidemiol. 2020 Apr 1;49(2):361-362e. doi: 10.1093/ije/dyz224. No abstract available. PMID 31725160
- [Background] Gideon N, Hawkes N, Mond J, Saunders R, Tchanturia K, Serpell L. Development and Psychometric Validation of the EDE-QS, a 12 Item Short Form of the Eating Disorder Examination Questionnaire (EDE-Q). PLoS One. 2016 May 3;11(5):e0152744. doi: 10.1371/journal.pone.0152744. eCollection 2016. PMID 27138364
- [Background] Morgan JF, Reid F, Lacey JH. The SCOFF questionnaire: a new screening tool for eating disorders. West J Med. 2000 Mar;172(3):164-5. doi: 10.1136/ewjm.172.3.164. No abstract available. PMID 18751246
- [Background] American Psychiatric Association D, Association AP. Diagnostic and statistical manual of mental disorders: DSM-5. American psychiatric association Washington, DC; 2013.
- [Background] Hill LS, Reid F, Morgan JF, Lacey JH. SCOFF, the development of an eating disorder screening questionnaire. Int J Eat Disord. 2010 May;43(4):344-51. doi: 10.1002/eat.20679. PMID 19343793
- Available data/document: Individual Participant Data Set — https://le.ac.uk/people/sam-tromans
- Available data/document: Study Protocol — https://le.ac.uk/people/sam-tromans
- Available data/document: Statistical Analysis Plan — https://le.ac.uk/people/sam-tromans
- Available data/document: Informed Consent Form — https://le.ac.uk/people/sam-tromans